CLINICAL TRIAL: NCT07276412
Title: Study on the Effect of a Health Education Programme Based on Gamification Strategies on Diet, Sedentary Behaviour and Daily Physical Activity in Primary School Children.
Brief Title: Study on the Effect of a Gamified Health Education Programme on Primary School Children
Acronym: BELLOTEX-SALUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Collaborators: Diputación Provincial de Badajoz (Unknown)
Responsible Party: Principal Investigator, Francisco Jose Rodriguez Velasco, Professor PhD, University of Extremadura, Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 32/2025
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Gamification in Health Education; Health Education
Keywords: school; child; obesity; physical activities; Health Education; Quality of Life; Gamification; sedentary
MeSH Terms: conditions — Health Education; Obesity; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): Group without weekly Health Education Programme and without reward for gamified activity
- Group A (Experimental): Group without weekly Health Education Programme and with reward for gamified activity
  Interventions: Behavioral: Intervention - A
- Group B (Experimental): Group with weekly Health Education Programme and no reward for gamified activity
  Interventions: Behavioral: Intervention - B
- Group C (Experimental): Group with weekly Health Education Programme and gamified activity rewards
  Interventions: Behavioral: Intervention - C

INTERVENTIONS:
Behavioral: Intervention - A — For this Intervention Group, rewards act as the main motivating factor for the children in this intervention group. Each time they complete the activities proposed in the application, they receive a "Bellotex Salud" avatar card, which symbolises their progress and identifies them as "Bellotex Masters". This gamified recognition boosts their involvement and reinforces their adherence to the intervention.
  In addition, this group does not attend weekly health education sessions, so the improvements observed can be attributed to the use of the app and the motivation generated by the rewards associated with the healthy habits worked on.
  Arms: Group A
Behavioral: Intervention - B — In this Intervention Group, participants will not have access to the rewards that act as the main motivating factor. Each time they complete the activities proposed in the application, they will pass the challenge but will not receive the "Bellotex Health" avatar card, which symbolises their progress and identifies them as "Bellotex Masters", thus allowing them to assess their potential involvement and adherence to the intervention without the reinforcement of gamified recognition.
  However, this group has access to weekly health education sessions, so the improvements observed can be attributed to the use of the app and the training received through these capsules associated with different healthy habits.
  Arms: Group B
Behavioral: Intervention - C — For this Intervention Group, rewards act as the main motivating factor. Each time they complete the activities proposed in the application, they receive a "Bellotex Salud" avatar card, which symbolises their progress and identifies them as "Bellotex Masters". This gamified recognition boosts their involvement and reinforces their adherence to the intervention.
  In addition, this group has access to weekly health education sessions, so that the improvements observed can be attributed to the use of the app and the training received through these capsules associated with different healthy habits.
  Arms: Group C

SUMMARY:
This randomised study evaluates the effectiveness of Health Education through a Gamified Health Programme on diet, sedentary behaviour and daily physical activity in primary school children.

DETAILED DESCRIPTION:
The prevalence of childhood obesity is high, being a serious health problem in our country, where 4 out of ten boys and girls are overweight.

Among the risk factors associated with obesity, the most prominent continue to be: lack of physical activity, those related to eating habits and excess time in front of screens.

Given that obesity is considered one of the most serious epidemics of the 21st century and that, if it is not stopped in childhood, it can cause serious health problems in adulthood, it is very important to work on this stage to reduce it.

In this evolutionary stage, children spend a lot of time in schools; Involving their teachers and teachers is important, but it is still necessary to do it with families as well. In this field, in that of fathers, mothers and/or guardians, the data shows parental weakness in aspects related to Health Education, such as those shown by the ALADINO 2019 study, where they point out that 7 out of 10 schoolchildren with excess weight are perceived by their parents as within a normal weight.

Our Health Education Program aims to ensure that the main actors (children) are accompanied and guided by their families and their teachers in the implementation of a series of activities associated with the achievement or improvement of daily habits. related to the previously indicated risk factors.

The Health Program, lasting 6 months, consists of daily, weekly or fortnightly activities. All of them interrelated and connected under the common objective of initiating or consolidating the aforementioned habits, in such a way that they improve the values of overweight in our sample.

We try to involve the child through gamification, through a story embodied in an interface that makes them feel involved. The achievement and fulfillment of each entrusted task will mean a series of achievements that will motivate the participants to continue accepting challenges.

ELIGIBILITY:
Inclusion Criteria:

* Pupils enrolled in primary education at schools in Extremadura.

Exclusion Criteria:

* All pupils diagnosed with special educational needs will be excluded.
* Pupils who join after the programme has started.
* Absence of informed consent signature to participate in the study and use of the BELLOTEX-SALUD application by the child's parents or legal guardians.
* Any condition that, in the opinion of the investigators, would disqualify the subject from participation in the study.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-07-24 (Estimated); Study Completion 2026-09-07 (Estimated)

PRIMARY OUTCOMES:
Changes in weekly physical activity at 12 weeks | 0 and 12 weeks
  Changes in time (minutes), distance (kilometres) and speed (km/h) measured by GPS through the BELLOTEX-SALUD application.
Changes in body fat mass composition over 12 weeks | 0 and 12 weeks
  Total patient body fat mass are measured as a kilogram (kg).
Changes in body weight composition over 12 weeks | 0 and 12 weeks
  Total patient weight are measured as a kilogram (kg).
Changes in Body Mass Index over 12 weeks | 0 and 12 weeks
  Weight (kg) and Height (m) will be combined to report BMI in kg/m^2.
Changes in the percentage of carbohydrates ingested over 12 weeks | 0 and 12 weeks
  A standardised food consumption questionnaire will be used to assess dietary habits, which collects food intake over 7 days. The weekly nutrient intake will be transformed into "Food Composition Tables". The value obtained will be the percentage of carbohydrates (%).
Changes in the percentage of fat ingested over 12 weeks | 0 and 12 weeks
  A standardised food consumption questionnaire will be used to assess dietary habits, which collects food intake over 7 days. The weekly nutrient intake will be transformed into "Food Composition Tables". The value obtained will be the percentage of fat ingested (%).
Changes in sedentary activity time over 12 weeks | 0 and 12 weeks
  Changes in "Screen-Time-Sedentary Behaviour Questionnaire" scores. The questionnaire consists of 23 items and assesses sedentary activity on weekdays and weekends.

SECONDARY OUTCOMES:
Changes in body fat-free mass composition over 12 weeks | 0 and 12 weeks
  Total patient body fat-free mass are measured as a kilogram (kg).
Changes in estimated total body water composition over 12 weeks | 0 and 12 weeks
  Total patient estimated total body water are measured as a kilogram (kg).
Changes in protein composition over 12 weeks | 0 and 12 weeks
  Total patient protein are measured as a kilogram (kg).
Changes in bone mineral composition over 12 weeks | 0 and 12 weeks
  Total patient bone mineral are measured as a kilogram (kg).
Changes in CUN-BAE index over 12 weeks | 0 and 12 weeks
  CUN-BAE are calculated as -44.988+(0.503×age) +(10.689 ×sex) +(3.172×BMI) -(0.026×BMI2) +(0.181×BMI×sex) -(0.02×BMI×age) -(0.005×BMI2 ×sex) +(0.00021×BMI2×age), where male=0 and female=1 for sex, measuring age in years.
Changes in phase angle bioimpedance over 12 weeks | 0 and 12 weeks
  Phase angle is measured in degrees (º).
Changes in the percentage of protein ingested over 12 weeks | 0 and 12 weeks
  A standardised food consumption questionnaire will be used to assess dietary habits, which collects food intake over 7 days. The weekly nutrient intake will be transformed into "Food Composition Tables". The value obtained will be the percentage of protein ingested (%).
Changes in the percentage of vitamins ingested over 12 weeks | 0 and 12 weeks
  A standardised food consumption questionnaire will be used to assess dietary habits, which collects food intake over 7 days. The weekly nutrient intake will be transformed into "Food Composition Tables". The value obtained will be the percentage of vitamins ingested (%).
Changes in kilocalorie intake over 12 weeks | 0 and 12 weeks
  A standardised food consumption questionnaire will be used to assess dietary habits, which collects food intake over 7 days. The weekly nutrient intake shall be transformed into "Food composition tables". The value obtained will be the number of kilocalories ingested (kcal).
Changes in adherence to the Mediterranean diet over 12 weeks | 0 and 12 weeks
  Changes in adherence to the Mediterranean diet. This will be studied using the KIDMED questionnaire, which consists of 16 items with values ranging from -1 (low adherence) to >1 (good adherence).
Changes in psychological parameters over 12 weeks | 0 and 12 weeks
  Changes in DAILY STRESS scores measured by the Inventory of Children's Daily Stress (IECI). The ICSI is a self-report questionnaire consisting of 22 items that assess the presence of daily stressors in children aged 6 to 12 years. The items are answered dichotomously (Yes/No) and are grouped into three subscales: Family, School, and Health/Psychosomatic, in addition to providing a total daily stress score. The direct scores reflect the number of stressful situations present for the child, with a possible total range of 0 to 22. There are no clinical cut-off points, but the scores are transformed into percentiles or T-scores adjusted for gender and school year, allowing the relative intensity of daily stress to be interpreted in comparison with the normative population.
Changes in digital connection time over 12 weeks | 0 and 12 weeks
  Weekly digital connection time (minutes) reported through the Bellotex-Salud app
Changes in quality of life indicators over 12 weeks | 0 and 12 weeks
  Changes in EQ-5D-Y-5L scores in children.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Extremadura, Badajoz, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No